CLINICAL TRIAL: NCT00275665
Title: A Phase III Multicenter Study of Valganciclovir for the Prevention of Late Cytomegalovirus Infection After Allogenic Hematopoietic Stem Cell Transplantation.
Brief Title: The Study is Being Done to See if Taking the Drug Valganciclovir Can Prevent CMV Infection.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Roche Pharma AG (Industry); Fred Hutchinson Cancer Center (Other); City of Hope National Medical Center (Other); University of Florida (Other); University of Michigan (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2124-01
Record Dates: First submitted 2006-01-10; First posted 2006-01-12 (Estimated); Last update posted 2011-12-19 (Estimated); Status verified 2011-12

CONDITIONS: Bone Marrow Stem Cell Transplant
MeSH Terms: interventions — Valganciclovir

INTERVENTIONS:
Drug: Valganciclovir

SUMMARY:
This study is being done in stem cell transplant recipients to see if taking the drug valganciclovir can prevent or reduce serious cytomegalovirus (CMV) infections that can occur 100 days or later after transplant.

DETAILED DESCRIPTION:
This study is a phase III, randomized, double-blind, palacebo-controlled, multicenter study of the drug valganciclovir. This study is to see if taking prophylactic doses of valganciclovir starting 100 days after stem cell transplantation can prevent late CMV from occurring.

Participants will be randomized (like a flip of a coin) into one of two groups. Neither the participant nor the doctor will know which group the participant is in. One group will receive the drug valganciclovir. The other group will receive a pill that looks like valganciclovir, but does not contain any active medicine (a placebo).

Participants enrolled in the study will take the drug by mouth daily starting at day 100 post stem cell transplant. Participants will also have blood samples taken along with their routine blood weekly, until day 270. Participants will also be required to return to their routine clinic visits.

Participants' acquiring an active CMV bloodstream infection at the time of the study will receive ganciclovir by the vein twice a day or a high dose of valganciclovir. Participants will be instructed to stop taking the study drug during the treatment time. After active CMV infection can no longer be detected, the treatment will be stopped. Patients will start taking the study drug and will be monitored for a CMV bloodstream infection until 270 days after transplant. Participants developing symptoms that look like CMV disease (pneumonia, infection of the intestines, eye infection) while on the study drug, will have an examination and lab tests to diagnose the organism. Participants that are hospitalized for CMV disease or for any other reason are asked to notify study personnel.

Participants will need to record study medicine taken in a daily study drug diary. Questionnaires will be filled out by the participant throughout the study, they will also be called monthly to see how they are doing and feeling overall.

After 270 days, participants will complete the study drug phrase. They will receive follow up phone calls on days 400, 520, and 640 days after transplant to see how they are doing.

ELIGIBILITY:
Participants who are undergoing allogeneic peripheral blood stem cell, cord blood, or marrow transplantation that are 18 years of age or older, may be eligible to participate in this study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2001-11; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
CMV disease
Invasive bacterial and fungal infections

SECONDARY OUTCOMES:
The occurrence of CMV infection or the occurrence of CMV disease (whichever occurs first) between enrollment and day 270 after transplantation.
Occurrence of CMV disease between randomization and day 270
The occurrence of other documented clinically significant human herpesvirus infections after randomization and day 270.
Survival to include a comparison of treatments at day 270 and day 640
Safety-comparison of adverse events and serious adverse events that occur on the two arms during the study

CONTACTS AND LOCATIONS:
Overall Officials: Mark R. Litzow, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States